CLINICAL TRIAL: NCT07030127
Title: A Phase 1, Participant- and Investigator-Blind, Randomized, Placebo-Controlled, Multiple-Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Multiple Subcutaneous Doses of LY3985863 in Healthy Chinese Participants
Brief Title: A Study of LY3985863 in Healthy Participants
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 27292; J4Z-MC-GIDH (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-06-12; First posted 2025-06-22 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- LY3985863 (Experimental): Administered subcutaneously (SC)
  Interventions: Drug: LY3985863
- Placebo (Placebo Comparator): Administered SC
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3985863 — Administered SC
  Arms: LY3985863
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate how well LY3985863 is tolerated and what side effects may occur in healthy Chinese participants. The study drug will be administered subcutaneously (SC) (under the skin).

Blood tests will be performed to investigate how the body processes the study drug and how the study drug affects the body.

ELIGIBILITY:
Inclusion Criteria:

* Are native Chinese participants
* Are overtly healthy
* Have body weight of at least 50.0 kilogram (kg) for male or 45.0 kg for female and a body mass index of 20.0 to 30.0 kilogram per square meter (kg/m²), inclusive
* Have a stable body weight within 3 months

Exclusion Criteria:

* Have known allergies to any components of the LY3985863 formulation
* Have concomitant disease known to influence skeletal muscle protein
* Have current or a history of comorbidities capable of significantly altering the absorption, metabolism, or elimination of drugs, of constituting a risk when taking the study medication or completing study procedures, or of interfering with the interpretation of the data
* Have a 12-lead echocardiogram (ECG) abnormality
* Have used within 3 months or intend to use medications during the study that promote weight loss

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-08-11 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with One or More Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline to Study Completion (Up to 19 Weeks)
  A summary of TEAEs and SAEs regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY3985863 | Predose on Day 1 up to Approximately Week 8 Post Dose
  PK: Cmax of LY3985863
PK: Area Under the Concentration Versus Time Curve (AUC) of LY3985863 | Predose on Day 1 up to Approximately Week 8 Post Dose
  PK: AUC of LY3985863

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No